CLINICAL TRIAL: NCT07030738
Title: Plant (Legumes) vs Animal-based (Meat) Protein Sources as an Anabolic and Metabolic-protective Options for Sarcopenic Obesity in Older Adults- A Randomized Controlled Trial
Brief Title: Plant vs Animal-based Protein Sources as an Anabolic and Metabolic-protective Options for SO in Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TLV-0540-23
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-05

CONDITIONS: Sarcopenic Obesity; Obesity and Obesity-related Medical Conditions; Obesity (Body Mass Index >30 kg/m2); Sarcopenia; Muscle Loss; Aging
Keywords: Plant-based diet; Red meat; Legumes; Protein intake; Anabolic diet; Resistance training; Muscle mass; Body composition; Older adults; Functional status; Sarcopenic obesity; Hypocaloric diet; Leucine; Physical function; Metabolic health; Aging population; Nutrition intervention; Randomized controlled trial
MeSH Terms: conditions — Obesity; Sarcopenia; Muscular Atrophy | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three parallel intervention arms: a legume-based high-protein hypocaloric diet (ProLegumes), a meat-based high-protein hypocaloric diet (ProMeat), or a mixed-source high-protein hypocaloric diet (ProMix). Each group follows their assigned intervention for the 12-week study period.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators, physical trainers, and outcomes assessors are blinded to group allocation. Participants and dietitians delivering the dietary intervention are not blinded, due to the nature of individualized nutrition counseling. All meals are coded neutrally to preserve blinding for trainers and assessors.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ProLegumes Diet (Experimental): Participants in this arm will follow a hypocaloric, high-protein diet primarily based on legumes as the main protein source. The diet aims to improve sarcopenic obesity outcomes over a 3-month intervention period, combined with home-based resistance training.
  Interventions: Behavioral: Legume-Based High-Protein Diet + Resistance Training
- ProMeat Diet (Active Comparator): Participants in this arm will follow a hypocaloric, high-protein diet primarily based on meat as the main protein source. This diet also aims to improve sarcopenic obesity outcomes over 3 months with the same exercise regimen.
  Interventions: Behavioral: Meat-Based High-Protein Diet + Resistance Training
- ProMix Diet (Active Comparator): Participants in this arm will follow a hypocaloric, high-protein diet that includes a combination of both legumes and meat as protein sources. The intervention period and exercise program are identical to the other arms.
  Interventions: Behavioral: Mixed Legume and Meat High-Protein Diet + Resistance Training

INTERVENTIONS:
Behavioral: Legume-Based High-Protein Diet + Resistance Training — Participants receive a hypocaloric, high-protein diet primarily based on legumes (e.g., lentils, beans, peas) designed to meet protein goals (~2g/kg body weight). Diet is combined with a structured home-based resistance training program performed 3 times per week for 12 weeks. The exercise includes progressive resistance exercises focusing on major muscle groups using body weight and resistance bands.
  Other Names: ProLegumes
  Arms: ProLegumes Diet
Behavioral: Meat-Based High-Protein Diet + Resistance Training — Participants follow a hypocaloric, high-protein diet emphasizing animal-based protein sources, mainly lean meats, to achieve ~2g/kg body weight protein intake. This dietary intervention is combined with a 12-week, home-based resistance training protocol, performed thrice weekly, targeting major muscle groups with progressive overload using body weight and resistance bands.
  Other Names: ProMeat
  Arms: ProMeat Diet
Behavioral: Mixed Legume and Meat High-Protein Diet + Resistance Training — Participants adhere to a hypocaloric, high-protein diet combining both legumes and lean meats as protein sources to reach ~2g/kg body weight. The dietary plan is paired with a 12-week home-based resistance training program, performed 3 times per week, emphasizing progressive resistance exercises for all major muscle groups using body weight and resistance bands.
  Other Names: ProMix
  Arms: ProMix Diet

SUMMARY:
This study is testing how different types of protein - from red meat, legumes (like lentils and beans), or a mix of both - affect muscle strength, body composition, and metabolic health in older adults with obesity who are also at risk for sarcopenia (loss of muscle mass and function). Participants will follow a personalized weight loss diet with one high-protein meal each day that includes either red meat, legumes, or both, along with a home-based strength training program. The study will last three months and will include health assessments such as blood tests, muscle and fat measurements, and physical function tests. The goal is to find out which type of protein source is most helpful for improving strength, reducing body fat, and supporting healthy aging.

ELIGIBILITY:
Inclusion Criteria:

* Aged 55 years or older.
* Diagnosed with obesity.
* At risk for sarcopenia, based on at least one of the following: Low score on the validated SARC-F-calf questionnaire (as suggested in prior studies). More than one comorbidity associated with sarcopenic obesity (e.g., diabetes, osteoporosis, cardiovascular disease, etc.). Polypharmacy: taking 8 or more prescribed medications. Evidence of strength or functional impairment, assessed using validated measurements at the baseline visit.

Exclusion Criteria:

* Recent use of steroid agents within the past 6 months (replacement therapy is allowed).
* Uncorrected hypothyroidism: TSH > 6 mIU/L.
* Diagnosis of malignancy within the past 5 years, except for non-melanoma skin cancer.
* Chronic kidney disease (CKD) at stage >1 (due to protein restriction needs).
* Recent (≤6 months) or unstable cardiovascular condition, or NYHA Class III or higher congestive heart failure.
* Currently performing resistance training.
* Currently undergoing nutritional therapy, have recently changed diet (<1 month), or are enrolled in active weight-loss programs or therapies (including lifestyle and/or pharmacotherapy). Note: Patients stable on GLP-1 agonists or other pharmacotherapy are eligible.
* Vegetarians/vegans, or individuals with aversion or allergy to all legumes or all red meat products.
* Habitual consumption of more than 3 servings/week of either legumes or red meat.
* Other medical, psychiatric conditions, or lab abnormalities that may pose a risk to participation.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
MetaboAnabolic Score | Baseline, Week 6, Week 12
  The MetaboAnabolic Score is a composite outcome designed to assess the intervention's efficacy in addressing sarcopenic obesity from both metabolic and functional perspectives. The score includes 10 variables: five metabolic (body fat percentage, intramuscular adipose tissue [IMAT], visceral fat area, blood pressure, and triglyceride or LDL levels) and five functional (leg muscle/lean mass, leg and arm strength, Timed Up and Go [TUG], and 2-minute walk test). A clinically meaningful threshold is defined for each variable based on scientific literature or expected changes from the hypocaloric intervention. One point is awarded for each variable that meets or exceeds the threshold, resulting in a total score ranging from 0 to 10. A higher score reflects greater overall improvement.

SECONDARY OUTCOMES:
Functional Performance Tests (TUG, STS, Gait, Strength) | Baseline, Week 6, Week 12
  TUG, 2-minute walk, 30s sit-to-stand, one-leg stand (gait, endurance, stability).
  Muscle strength of upper and lower limbs measured via handheld dynamometers. Gait variability and balance measured using Mobility Lab (OPAL) sensors
C-Reactive Protein (CRP) Levels | Baseline, Week 6, Week 12
  High-sensitivity CRP will be measured via blood samples to assess systemic inflammation. CRP is a biomarker associated with metabolic and cardiovascular risk.
Lipid Profile (Triglycerides, LDL, HDL, Total Cholesterol) | Baseline, Week 6, Week 12
  Fasting blood samples will be used to assess lipid parameters including triglycerides, low-density lipoprotein (LDL), high-density lipoprotein (HDL), and total cholesterol. These are key indicators of cardiovascular and metabolic health. Changes will be compared between intervention groups.
Glycemic Control (Fasting Glucose, Insulin, HOMA-IR) | Baseline, Week 6, Week 12
  Fasting glucose and insulin levels will be used to evaluate glycemic control and insulin sensitivity. Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) will be calculated.
Resting Metabolic Rate (RMR) | Baseline and Week 12
  RMR will be measured via indirect calorimetry under standardized fasting and resting conditions. It reflects basal energy expenditure and can indicate metabolic adaptation or dysfunction. Changes will be analyzed in the context of body composition shifts.
Body Composition (Lean Mass, Fat Mass, Visceral Fat Area) | Baseline, Week 6, Week 12
  Dual-energy X-ray absorptiometry (DXA) and bioelectrical impedance analysis will be used to assess lean body mass, total fat mass, and visceral fat area. Changes in these components will provide insight into the impact of the dietary interventions on sarcopenic obesity.
Muscle Quality Indices (Glycogen and Intramuscular Fat Levels) | Baseline, Week 6, Week 12
  Quantitative ultrasound will assess skeletal muscle glycogen storage and intramuscular fat infiltration (IMAT). This will be assessed by ultrasound of rectus femoris with MuscleSound® software, which analyzes cross-sectional area, thickness, and composition. These indices serve as biomarkers of muscle health and metabolic quality, with changes reflecting diet and exercise response.
Ambulatory Blood Pressure (24-hour monitoring) | Baseline, Week 6, Week 12
  Blood pressure will be monitored over 24 hours using a validated automatic ambulatory device to capture daily fluctuations.
Quality of Life (SF-12) | Baseline, Week 6, Week 12
  Health-related quality of life assessed using the validated SF-12 questionnaire, translated and culturally adapted to Hebrew.
Hormonal Markers (Testosterone, IGF-1, Vitamin D) | Baseline, Week 6, Week 12
  Serum levels of testosterone (bioavailable and free), IGF-1, and 25-hydroxyvitamin D will be measured using standard clinical protocols.

OTHER OUTCOMES:
Banked Blood and Serum for Future Biomarker and Epigenetic Analysis | Baseline, Week 6, Week 12
  Frozen plasma and blood samples will be collected and stored at -20 °C and - 80 °C respectively for future testing of myokines, adipokines, and epigenetic markers.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Tel Aviv, Israel